CLINICAL TRIAL: NCT01159574
Title: A Phase II Study of Dexamethasone (DECADRON®), Clarithromycin (BIAXIN®), and Pomalidomide (CC-4047®) for Subjects With Relapsed or Refractory Multiple Myeloma
Brief Title: Study of Decadron, Biaxin, and Pomalidomide in Relapsed/Refractory Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1004011012; PO-MM-PI-0023 (Other Grant/Funding Number: Celgene)
Record Dates: First submitted 2010-06-16; First posted 2010-07-09 (Estimated); Results first posted 2017-04-12 (Actual); Last update posted 2019-06-11 (Actual); Status verified 2019-05

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Dexamethasone; Calcium Dobesilate; Clarithromycin; pomalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- all patients (Experimental): ClaPd therapy:
  Dexamethasone (40mg ) will be given on days 1, 8, 15, 22 of a 28-day cycle. Clarithromycin (Biaxin®) will be given orally at a dose of 500 mg twice a day on days 1-28 of a 28 day cycle.
  Pomalidomide will be given 4mg daily for days 1-21 of each 28 day cycle. Dosing will be in the morning at approximately the same time each day.
  Interventions: Drug: dexamethasone; Drug: clarithromycin; Drug: Pomalidomide

INTERVENTIONS:
Drug: dexamethasone — 40mg will be given on days 1, 8, 15, 22 of a 28-day cycle
  Other Names: Decadron
Drug: clarithromycin — orally at a dose of 500 mg twice a day on days 1-28 of a 28 day cycle
  Other Names: Biaxin
Drug: Pomalidomide — orally 4mg daily for days 1-21 of each 28 day cycle
  Other Names: CC-4047

SUMMARY:
This study is intended to investigate the combination of the combination of dexamethasone (Decadron®), Clarithromycin (Biaxin®), and pomalidomide (CC-4047®) [ClaPd] in multiple myeloma patients who have relapsed or refractory disease who have failed prior treatment with lenalidomide when used alone or in combination with corticosteroids. Primary endpoint will be response rate to treatment. Secondary endpoints will include toxicity of the combination, time to maximum response, and time to disease progression

DETAILED DESCRIPTION:
This phase II study is a treatment program for patients with relapsed or refractory multiple myeloma who have had prior treatment with lenalidomide. Up to 54 patients will be enrolled. Patients who sign informed consent form and fulfill all eligibility criteria will be enrolled.

ClaPd therapy:

Dexamethasone (40mg ) on days 1, 8, 15, 22 of a 28-day cycle. Clarithromycin given orally at a dose of 500 mg twice a day on days 1-28 of a 28 day cycle.

Pomalidomide will be given 4mg daily for days 1-21 of each 28 day cycle.

Serial clinic visits and laboratory measurements will be performed to monitor for treatment response. Those patients who demonstrate progression of disease at any point during ClaPd therapy will be taken off study.

At the end of every cycle (which may coincide with day 1 of the new cycle), response and toxicity will be evaluated. During cycle 1, patients will have labwork done weekly (CBC with differential and blood electrolytes). All patients will remain on study until disease progression or side effects become excessive. Patients who achieve a stable plateau may be taken off study if eligible to proceed to high dose chemotherapy and autologous stem cell transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Subject must voluntarily sign and understand written informed consent.
* Age > 18 years at the time of signing the consent form.
* Histologically confirmed MM
* Relapsed or refractory myeloma, progression of disease either after prior therapy or lack of response to currently used therapy.
* Relapsed or progressive disease after at least 3 prior therapeutic treatments or regimens for multiple myeloma.
* Must have been previously treated with lenalidomide and has been determined to be refractory, resistant, or relapsed.
* Measurable disease as defined by > 0.5 g/dL serum monoclonal protein, >0.1 g/dL serum free light chains, >0.2 g/24 hrs urinary M-protein excretion, and/or measurable plasmacytoma(s).
* Karnofsky performance status ≥70% (>60% if due to bony involvement of myeloma
* Females of childbearing potential (FCBP)† must have a negative serum or urine pregnancy test with a sensitivity of at least 50 mIU/mL within 10 - 14 days prior to and again within 24 hours of prescribing lenalidomide and thalidomide (prescriptions must be filled within 7 days) and must either commit to continued abstinence from heterosexual intercourse or begin TWO acceptable methods of birth control, one highly effective method and one additional effective method AT THE SAME TIME, at least 4 weeks before she starts taking lenalidomide. FCBP must also agree to ongoing pregnancy testing. Men must agree to use a latex condom during sexual contact with females of child bearing potential even if they have had a successful vasectomy. See Appendix V: Pomalidomide Risks of Fetal Exposure, Pregnancy Testing Guidelines and Acceptable Birth Control Methods. †A female of childbearing potential is a sexually mature woman who: 1) has not undergone a hysterectomy or bilateral oophorectomy; or 2) has not been naturally postmenopausal for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months).
* Able to take aspirin daily as prophylactic anticoagulation (patients intolerant to ASA may use warfarin or low molecular weight heparin). †
* 1ife expectancy ≥ 3 months
* Subjects must meet the following laboratory parameters:

Absolute neutrophil count (ANC) ≥750 cells/mm3 (1.0 x 109/L) Platelets count ≥ 50,000/mm3 (75 x 109/L) Serum SGOT/AST ≤ 2.0 x upper limits of normal Serum SGPT/ALT <3.0 x upper limits of normal (ULN) Serum creatinine ≤ 2.5 x upper limits of normal Serum total bilirubin ≤ 1.5 x upper limits of normal

Exclusion Criteria:

* Patients with non-secretory MM (no measurable monoclonal protein, free light chains, and/or M-spike in blood or urine).
* Prior history of other malignancies (except for basal cell or squamous cell carcinoma of the skin or carcinoma in situ of the cervix or breast) unless disease free for ≥ 5 years.
* Myocardial infarction within 6 months prior to enrollment, or NYHA(New York Hospital Association) Class III or IV heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias, electrocardiographic evidence of acute ischemia or active conduction system abnormalities.
* Known HIV infection
* Known hepatitis B or hepatitis C infection.
* Active viral or bacterial infections or any coexisting medical problem that would significantly increase the risks of this treatment program.
* Any coexisting medical problem or laboratory evaluation that, in the treating physician's or principal investigator's opinion, makes the patient unsuitable to participate in this clinical trial.
* Known hypersensitivity to thalidomide or lenalidomide.
* History of thromboembolic event within the past 6 months prior to enrollment.
* Any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from signing the informed consent form.
* Pregnant or breast feeding females.
* Any condition, including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study.
* Use of any other experimental drug or therapy within 14 days of baseline.
* Known hypersensitivity to thalidomide or lenalidomide.
* The development of erythema nodorum if characterized by a desquamating rash while taking thalidomide, CC-4047 or similar drugs.
* Any prior use of CC-4047.
* Concurrent use of other anti-cancer agents or treatments.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2010-08 (Actual); Primary Completion 2015-05-05 (Actual); Study Completion 2015-05-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ruben Niesvizky, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medical College, New York, New York, United States

REFERENCES:
- [Derived] Mark TM, Forsberg PA, Rossi AC, Pearse RN, Pekle KA, Perry A, Boyer A, Tegnestam L, Jayabalan D, Coleman M, Niesvizky R. Phase 2 study of clarithromycin, pomalidomide, and dexamethasone in relapsed or refractory multiple myeloma. Blood Adv. 2019 Feb 26;3(4):603-611. doi: 10.1182/bloodadvances.2018028027. PMID 30792190

RESULTS

PARTICIPANT FLOW:
Groups:
- All Patients: ClaPd therapy:
  Dexamethasone (40mg ) will be given on days 1, 8, 15, 22 of a 28-day cycle. Clarithromycin (Biaxin®) will be given orally at a dose of 500 mg twice a day on days 1-28 of a 28 day cycle.
  Pomalidomide will be given 4mg daily for days 1-21 of each 28 day cycle. Dosing will be in the morning at approximately the same time each day.
  dexamethasone: 40mg will be given on days 1, 8, 15, 22 of a 28-day cycle
  clarithromycin: orally at a dose of 500 mg twice a day on days 1-28 of a 28 day cycle
  Pomalidomide: orally 4mg daily for days 1-21 of each 28 day cycle
Period: Treatment Phase
Arm/Group | All Patients
Started | 121
Completed (Completion defined as those that were removed from treatment due to disease progression.) | 100
Not Completed | 21
Not completed — non-evaluable/not included in analysis | 1
Not completed — Adverse Event | 3
Not completed — Death | 6
Not completed — Physician Decision | 2
Not completed — Withdrawal by Subject | 7
Not completed — still on treatment | 2
Period: Follow Up Phase
Arm/Group | All Patients
Started (Follow-up includes all patients except those that passed away on treatment or were non-evaluable.) | 112
Completed | 92 (Completion defined as those that are no longer in long term follow up due to death.)
Not Completed | 20
Not completed — Lost to Follow-up | 2
Not completed — still being followed for overall surviva | 18

BASELINE CHARACTERISTICS:
Population: 121 subject signed consent; 1 subject was not considered to be evaluable and was not included in any analysis.
Arm/Group | All Patients
Number analyzed (Participants) | 120
Age, Continuous [Median (Full Range); unit: years] | 63 [42 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 62
  Male | 58
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6
  Not Hispanic or Latino | 112
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 8
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 12
  White | 93
  More than one race | 0
  Unknown or Not Reported | 7
Hemoglobin [Median (Full Range); unit: g/dL] | 10.4 [6.4 to 14.6]
Range of Prior Therapies [Median (Full Range); unit: years] | 5 [3 to 15]
Beta-2 microglobulin at baseline (in mg/L) [Median (Full Range); unit: mg/L] | 35 [1.2 to 40.4]
lactage dehydrogenase at baseline (U/L) [Median (Full Range); unit: u/l] | 170.5 [79 to 1353]

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate
Description: Best response rate was recorded for all patients, using the IMWG criteria.
Time Frame: from baseline to cycle with maximum response, which was achieved on average after 2 cycles
Measure: Count of Participants; unit: Participants
Arm/Group | All Patients
Number analyzed (Participants) | 120
Participants
  stringent Complete Response | 6
  Complete Response | 1
  Very Good Partial Response | 20
  Partial Response | 43
  Minimal Response | 8
  stable disease | 29
  Not evaluable | 3
  progression of disease | 10

2. Secondary Outcome: Time to Maximum Response, Expressed as Number of Cycles of Treatment to Maximum Response
Time Frame: From baseline to cycle of maximum response, which occurred on average after 2 cycles; 1 cycle = 28 days
Measure: Mean (Full Range); unit: cycles
Arm/Group | All Patients
Number analyzed (Participants) | 120
cycles | 2.19 [1 to 18]

3. Secondary Outcome: Time to Disease Progression (Progression Free Survival)
Time Frame: From start of treatment, to date of disease progression
Population: 18 patients were removed from study for reasons other then disease progression; 2 patients are still receiving treatment.
Measure: Mean (Full Range); unit: days
Arm/Group | All Patients
Number analyzed (Participants) | 100
days | 272 [21 to 1430]

ADVERSE EVENTS:
Time Frame: Adverse events were recorded from baseline until removal from study. Serious adverse events were recorded from baseline until 30 days after the last dose of study drug.
Description: Adverse events were recorded using the CTCAE version 4.0. The adverse events listed includes serious adverse events. Serious adverse events were recorded from baseline unti
Arm/Group | All Patients
Serious Adverse Events (participants affected / at risk) | 59/120
Other Adverse Events (participants affected / at risk) | 120/120
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Patients (N=120)
acute renal failure (Renal and urinary disorders) | 1 (1)
agitation (Psychiatric disorders) | 1 (1)
altered mental status (Psychiatric disorders) | 1 (1)
anemia (Blood and lymphatic system disorders) | 3 (3)
atrial fibrillation (Cardiac disorders) | 1 (1)
back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
behavior changes (Psychiatric disorders) | 1 (1)
bowel obstruction (Gastrointestinal disorders) | 1 (1)
cellulitis (Infections and infestations) | 1 (1)
chest pain (Musculoskeletal and connective tissue disorders) | 1 (1)
chronic kidney insufficiency (Renal and urinary disorders) | 1 (1)
complications of MM (leading to death) (Investigations) | 1 (1)
confusion (Psychiatric disorders) | 2 (3)
cough (Infections and infestations) | 1 (1)
creatinine increased (Metabolism and nutrition disorders) | 1 (1)
death (General disorders) | 1 (1)
dehydration (Metabolism and nutrition disorders) | 6 (6)
diarrhea (Gastrointestinal disorders) | 5 (5)
diffuse small bowl ileus (Gastrointestinal disorders) | 1 (1)
diverticullitis (Infections and infestations) | 1 (1)
dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (3)
epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
fall (General disorders) | 1 (1)
fatigue (General disorders) | 1 (1)
febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
fever (Infections and infestations) | 4 (4)
fracture (Musculoskeletal and connective tissue disorders) | 4 (4)
gastroenteritis (Infections and infestations) | 1 (1)
hypotension (Vascular disorders) | 3 (3)
hallunication (Psychiatric disorders) | 1 (1)
pain (hip, rib) (Musculoskeletal and connective tissue disorders) | 1 (1)
pain (rib) (Musculoskeletal and connective tissue disorders) | 1 (1)
hypercalcemia (Metabolism and nutrition disorders) | 1 (1)
hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
hyperkalemia (Metabolism and nutrition disorders) | 1 (1)
infection (Infections and infestations) | 1 (1)
intrcranial bleed (Investigations) | 1 (1)
lower back pain (Musculoskeletal and connective tissue disorders) | 2 (2)
lung infection (Infections and infestations) | 15 (16)
muscle weakness (Musculoskeletal and connective tissue disorders) | 2 (2)
nausea (Gastrointestinal disorders) | 2 (2)
neutropenia (Blood and lymphatic system disorders) | 3 (3)
neutropenic fever (Infections and infestations) | 4 (4)
pancytopenia (Blood and lymphatic system disorders) | 1 (1)
parainfluenza virus infection (Infections and infestations) | 1 (1)
pulmonary emboli (Respiratory, thoracic and mediastinal disorders) | 1 (1)
rash (Skin and subcutaneous tissue disorders) | 1 (1)
renal insufficiency (Infections and infestations) | 4 (4)
rhinovirus (Infections and infestations) | 1 (1)
sepsis (Infections and infestations) | 3 (3)
skin infection (including cellulitis) (Infections and infestations) | 3 (4)
suspected seizure (Nervous system disorders) | 1 (1)
syncopal episode (Psychiatric disorders) | 2 (2)
thrombocytopenia (Blood and lymphatic system disorders) | 2 (2)
thromboembolic event (Vascular disorders) | 2 (2)
transient word finding difficulity (General disorders) | 1 (1)
vomiting (Gastrointestinal disorders) | 5 (5)
weakness (including associated pain/tiredness) (General disorders) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | All Patients (N=120)
neuro mood (Nervous system disorders) | 6
psychomotor agitation (Nervous system disorders) | 6
bone pain (Musculoskeletal and connective tissue disorders) | 6
renal failure/insufficiency (Renal and urinary disorders) | 6
epistaxis (Respiratory, thoracic and mediastinal disorders) | 6
Skin Infection (Infections and infestations) | 6
Thrush (Infections and infestations) | 6
cramping (Gastrointestinal disorders) | 7
dry mouth (Gastrointestinal disorders) | 7
confusion (Nervous system disorders) | 7
Lower extremity DVT (Vascular disorders) | 7
chest pain (muscular) (Musculoskeletal and connective tissue disorders) | 7
cushingoid (Skin and subcutaneous tissue disorders) | 7
UTI (Infections and infestations) | 7
dehydration (Gastrointestinal disorders) | 8
hypermagnesemia (Metabolism and nutrition disorders) | 8
hypernatremia (Metabolism and nutrition disorders) | 8
agitation (Nervous system disorders) | 8
Paresthesia (Nervous system disorders) | 8
rash maculo papular (Skin and subcutaneous tissue disorders) | 8
hoarseness (Respiratory, thoracic and mediastinal disorders) | 8
postnasal drip (Respiratory, thoracic and mediastinal disorders) | 8
Pneumonia (Infections and infestations) | 8
bruising (Vascular disorders) | 9
Hyperuricemia (Renal and urinary disorders) | 9
hypercalcemia (Metabolism and nutrition disorders) | 10
weight gain (Metabolism and nutrition disorders) | 10
facial flushing (Skin and subcutaneous tissue disorders) | 10
hyperhidrosis (Skin and subcutaneous tissue disorders) | 10
fall (General disorders) | 10
weight loss (Metabolism and nutrition disorders) | 11
pain in general (Musculoskeletal and connective tissue disorders) | 11
pain in legs (Musculoskeletal and connective tissue disorders) | 11
nasal congestion (Respiratory, thoracic and mediastinal disorders) | 11
sore throat (Infections and infestations) | 11
bloating (Gastrointestinal disorders) | 12
CKD (Renal and urinary disorders) | 12
abdominal pain/discomfort (Gastrointestinal disorders) | 13
flatulance (Gastrointestinal disorders) | 13
generalized weakness (General disorders) | 13
fever (Infections and infestations) | 13
hyperkalemia (Metabolism and nutrition disorders) | 14
headache (Nervous system disorders) | 14
hip pain (Musculoskeletal and connective tissue disorders) | 14
vomiting (Gastrointestinal disorders) | 15
rib pain (Musculoskeletal and connective tissue disorders) | 15
rash (Skin and subcutaneous tissue disorders) | 15
anorexia (Metabolism and nutrition disorders) | 17
anxiety/stress (Nervous system disorders) | 17
dyspepsia (Gastrointestinal disorders) | 18
shoulder pain (Musculoskeletal and connective tissue disorders) | 18
blurry vision (Eye disorders) | 18
elevated AST (Metabolism and nutrition disorders) | 19
depression (Nervous system disorders) | 19
dysgeusia (Nervous system disorders) | 19
lung infection (Infections and infestations) | 19
muscle spasms/cramps (Musculoskeletal and connective tissue disorders) | 22
nausea (Gastrointestinal disorders) | 23
Hyperbilirubinemia (Metabolism and nutrition disorders) | 23
Hypokalemia (Metabolism and nutrition disorders) | 23
cough (Infections and infestations) | 24
dizziness / lightheaded (Nervous system disorders) | 25
URI (Infections and infestations) | 27
tremor (Nervous system disorders) | 29
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 30
Hypophosphatemia (Metabolism and nutrition disorders) | 31
constipation (Gastrointestinal disorders) | 32
muscle weakness (Musculoskeletal and connective tissue disorders) | 33
elevated ALT (Metabolism and nutrition disorders) | 36
elevated ALK (Metabolism and nutrition disorders) | 36
insomnia (General disorders) | 36
peripheral neuropathy (Nervous system disorders) | 37
edema (Vascular disorders) | 38
back pain (Musculoskeletal and connective tissue disorders) | 39
diarrhea (Gastrointestinal disorders) | 44
increased creatinine (Metabolism and nutrition disorders) | 46
Hypomagnesemia (Metabolism and nutrition disorders) | 51
hyponatremia (Metabolism and nutrition disorders) | 62
hypocalcemia (Metabolism and nutrition disorders) | 66
Hypoalbuminemia (Metabolism and nutrition disorders) | 70
hypoglycemia (Metabolism and nutrition disorders) | 73
Anemia (Blood and lymphatic system disorders) | 74
fatigue (General disorders) | 75
hyperglycemia (Metabolism and nutrition disorders) | 77
Thrombocytopenia (Blood and lymphatic system disorders) | 85
Leukopenia (Blood and lymphatic system disorders) | 86
Lymphopenia (Blood and lymphatic system disorders) | 89
Neutropenia (Blood and lymphatic system disorders) | 99

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less